CLINICAL TRIAL: NCT03190486
Title: Perception of Baby's Painful Cry: Investigation in fMRI to Neuronal Activity Related to Empathy in Adults
Brief Title: Perception of Baby's Painful Cry in fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University Hospital of Saint-Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1708071; ID-RCB (Other: 2017-A01180-53)
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Magnetic Resonance Imaging; Neuronal Activity
Keywords: Baby cries; pain; brain responses; neuroimaging; fMRI
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: 20 men and 20 women : group "non parent" 20 father and 20 mother : group "parent"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Men contact-less with children (Experimental): functional Magnetic Resonance Imaging (fMRI).
  Interventions: Other: functional Magnetic Resonance Imaging (fMRI)
- Women contact-less with children (Experimental): functional Magnetic Resonance Imaging (fMRI).
  Interventions: Other: functional Magnetic Resonance Imaging (fMRI)
- Father contact-less with children (Experimental): functional Magnetic Resonance Imaging (fMRI).
  Interventions: Other: functional Magnetic Resonance Imaging (fMRI)
- Mother contact-less with children (Experimental): functional Magnetic Resonance Imaging (fMRI).
  Interventions: Other: functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Other: functional Magnetic Resonance Imaging (fMRI) — During fMRI, healthy volunteers will listen 80 baby's cry.
  Other Names: fMRI

SUMMARY:
Crying is the primary signaling strategy available to the human newborn for eliciting parental care. Yet, the investigators only have superficial understanding of the information carried by cries, and how this information is perceived by parents. Using modern tools of sound processing and functional Magnetic Resonance Imaging (fMRI) experiment, this study aims to investigate cry-induced brain activation in adult depending on the cry's acoustic properties expressing various degrees of stress and distress levels. For that, Adults will be tested inside a fMRI magnet to determine their brain activations elicited by different babies cries according to whether the cry was evoked in a pain situation or not. The cerebral activity will be investigated in relation to acoustic features of cries (e.g. with pitch and/or roughness variations). To test if the gender or parentally of adult listeners influence their perceptions and brain responses, the task will be applied to 2 different groups (men and women not-parents). The hypothesis is that the brain of adult listeners will be able to discriminate adequately the intensity of the pain mediated by the cries. This process should involve brain areas such as the insular and the orbito frontal cortex that are known to participate in the integration of pain intensity and pain controls. The experiment should also determine which one of the acoustic features is able to transmit pain and to recruit brain areas involved in pain processes.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged between 18 and 50
* Contact-less with children
* right-handed
* Giving their written informed consent
* Subject who agreed to communicate MRI results to their attending physician
* French Social Security affiliation

Exclusion Criteria:

* any contraindications to pass an fMRI test
* Pregnant woman

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 40 women and 40 men
Enrollment: 80 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
BOLD (blood-oxygen-level dependent) -contrast imaging | at inclusion
  Measure of blood-oxygen-level dependent with fMRI during listening to natural crying.

SECONDARY OUTCOMES:
BOLD (blood-oxygen-level dependent) -contrast imaging | at inclusion
  Measure of blood-oxygen-level dependent with by fMRI during listening to artificial crying.
impact of gender and parenting on perception of baby's cry | at inclusion
  Measure of blood-oxygen-level dependent with by fMRI during listening to artificial crying.

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Service de Neurologie - CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fauchon C, Corvin S, Faillenot I, Patural H, Reby D, Peyron R, Mathevon N. Parenting and empathy capabilities drive brain response to pain cues in baby cries. Pain. 2026 Jan 15. doi: 10.1097/j.pain.0000000000003914. Online ahead of print. PMID 41557145